CLINICAL TRIAL: NCT04780204
Title: A Multicenter, Open-label, Single Arm Trial for the Effectiveness of Antiviral Treatment in Cirrhotic Patients with Low-level Hepatitis B Virus DNA Levels with a Comparison to Matched Historical Controls (ATTACH)
Brief Title: Effectiveness of Antiviral Treatment in Cirrhotic Patients with Low-level Hepatitis B Virus DNA Levels
Acronym: ATTACH
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government)
Responsible Party: Principal Investigator, Young-Suk Lim, PhD, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-KR-320-6132
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Therapeutics; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antiviral Treatment (Experimental): Tenofovir Alafenamide 25mg once daily , Oral
  Interventions: Drug: Treatment
- Matched Historical Controls (No Intervention): Patients who did not receive antiviral treatment during their follow-up period, and matched with the treatment group in a 1:2 ratio according to their baseline characteristics

INTERVENTIONS:
Drug: Treatment — Tenofovir Alafenamide 25 mg oral once daily
  Other Names: Tenofovir alafenamide
  Arms: Antiviral Treatment

SUMMARY:
Multicenter, Open-label, Single arm Trial with Matched Historical controls. Male and female adults with compensated liver cirrhosis due to chronic hepatitis B virus infection who have low-level viremia.

To assess the efficacy of Tenofovir Alafenamide (TAF) in reducing liver-related events (hepatocellular carcinoma, liver-related events and death, decompensated liver cirrhosis) in cirrhotic chronic hepatitis B patients with low-level viremia compared with matched historical controls.

DETAILED DESCRIPTION:
1. This clinical trial is a multicenter, open label, single arm study in cirrhotic chronic hepatitis B patients with low-level viremia.
2. Approximately 200 subjects meeting eligibility criteria will be enrolled and randomized (1:2) to Treatment Arm (A) or , Matched Historical Controls Arm (B), as below:

   * Treatment Arm (A): 200 subjects, TAF 25mg once daily with food for 3 years
   * Matched Historical Controls Arm (B): 400 subjects, patients who did not receive antiviral treatment during their follow-up period, and matched with the treatment group in a 1:1 ratio according to their baseline characteristics
3. Treatment Arm is scheduled to be followed up to 3 years.

The analysis population of this study consists of the Full Analysis Set (FAS), which can evaluate efficacy. The treatment group includes patients who received any dose of study medication (TAF), while the control group consists of patients who did not receive antiviral treatment and were matched by propensity score (PS) from those under observation. Unless otherwise specified, the FAS will be used for primary and secondary efficacy endpoints.

Statistical analyses for the primary efficacy endpoint will be performed at a two-sided significance level of 5%, aligned with the sample size calculation.

PS will be estimated using logistic regression, incorporating variables such as age, gender, HBeAg positivity, HBV DNA level, ALT, platelet count, albumin, total bilirubin, creatinine, prothrombin time, diabetes, hypertension, and family history of hepatocellular carcinoma. The groups will be matched 1:2 using nearest neighbor matching. Baseline characteristics between the matched groups will be compared using standardized mean difference (SMD), with an absolute SMD <0.1 indicating good balance.

The 3-year cumulative incidence of the primary endpoint will be estimated using the Kaplan-Meier method. For comparisons between PS-matched groups, a Cox proportional hazards model with robust variance estimation will be used to account for matching, reporting HR and 95% confidence intervals.

For hepatocellular carcinoma incidence, mortality, liver transplantation, decompensated liver function (Child-Pugh score ≥8), and cirrhosis-related complications, 1-, 2-, and 3-year incidence rates will be estimated with Kaplan-Meier. Cox models with robust variance will be used for group comparisons, reporting HR and 95% confidence intervals.

HBsAg loss and viral response (HBV DNA <15 IU/mL) are binary outcomes, summarized by frequency and proportion in each group. Comparisons will be made using a Poisson regression model with Generalized Estimating Equations (GEE), reporting relative risk (RR) and 95% confidence intervals.

Fibroscan changes, treatment response, duration, and health-related quality of life by disease status (hepatitis, cirrhosis, hepatocellular carcinoma) will be analyzed using GEE, accounting for the matched-pair design.

In the PS-matched retrospective control group, the 1-, 2-, and 3-year cumulative probabilities of initiating antiviral therapy due to serum HBV DNA ≥2,000 IU/mL will be estimated via Kaplan-Meier.

Two official analyses will be conducted: an interim analysis (using data collected by October 2024) and a final analysis. No correction for type 1 error inflation from multiple testing will be applied in the interim analysis.

For sensitivity analysis, multivariable analyses will be performed using the unmatched dataset for primary and secondary endpoints. Depending on outcome type, Cox models and Poisson regression will be employed, using the covariates from the PS estimation for adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to study entry
2. Age ≥30 years and ≤80 years at the time of screening
3. Chronic hepatitis B infection defined as HBsAg (+) or HBV DNA (+) for at least 6 months prior to the Screening visit, or medical records indication a chronic hepatitis B virus infection by meeting all of the following criteria at the time of screening. (1) HBsAg (+), (2) HBV DNA (+), and (3) HBcAb IgM (-)
4. Either HBeAg (+) or HBeAg (-)
5. Serum HBV DNA levels ≥20 IU/mL and <2,000 IU/mL at the time of screening
6. Evidence of liver cirrhosis defined as meeting any of the following criteria:

   * Radiological evidence of liver cirrhosis by ultrasound, CT, or MRI
   * Platelet count <150,000 /mm3
   * Presence of esophageal or gastric varices by endoscopy in 2 years before the timing of screening
   * Clinically significant portal hypertension
   * Fibroscan ≥12.0 kPa (if the test was done in 6 months before the time of screening)
7. Estimated creatinine clearance ≥30 ml/min (by calculation of creatinine clearance or using the CKD-EPI equation)
8. Ability to comply with all study requirements

Exclusion Criteria:

1. Confirmed known co-infection with HCV, HIV, or HDV
2. Current alcohol (60g/day) or substance abuse judged by the investigator that will potentially interfere with subject compliance
3. Any history of, or current evidence of, clinical hepatic decompensation (e.g., ascites, encephalopathy, variceal hemorrhage, or Child-Pugh score of ≥8, with the exception of Gilbert syndrome) in 1 year before the time of screening
4. Currently on or have received therapy with Interferon or immunosuppressant (including systemic chemotherapy) within 12 months prior to the screening
5. Requirement for chronic use of systemic immunosuppressant including, but not limited to, corticosteroid (prednisone equivalent of >40 mg/day for >2 weeks), azathioprine, or monoclonal antibodies
6. Received solid organ or bone marrow transplant
7. History of severe, life-threatening or other significant sensitivity to any excipients of the study drugs
8. Any other clinical conditions (cardiovascular, respiratory, neurologic, or renal conditions) or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.
9. Currently on or have received antiviral treatment for ≥ 2 weeks within 6 months prior to the screening
10. History or current evidence of hepatocellular carcinoma (HCC), or high α-fetoprotein (AFP) > 20 ng/mL. But, the patients with AFP > 20 ng/mL can be enrolled if AFP shows decreasing trend and there is no evidence of HCC by dynamic CT or MRI)
11. Malignancy other than hepatocellular carcinoma within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (within 2 years prior to screening with confirmation of no evidence of disease). Subjects under evaluation for possible malignancy are not eligible.
12. Concurrent enrollment in another clinical study for other type of antiviral treatment for CHB or immune modulatory drug within 3 months prior to randomization, participation to an observational (non-interventional) clinical studies or interventional studies not using anti-HBV or immune modulatory drugs, or during the follow-up period of an interventional study are not exclusion criteria.
13. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of composite clinical events | From randomization the composite clinical events will be collected every 6weeks , assessed up to 36months
  hepatocellular carcinoma, death, liver transplantation, decompensated liver cirrhosis defined as Child-Pugh score ≥8, liver cirrhosis-related complications,liver-related unexpected hospital admission

SECONDARY OUTCOMES:
Cumulative incidence | From randomization the composite clinical events will be collected every 1year , assessed up to 3years
  Death, hepatocellular carcinoma , Liver transplantation, decompensated liver cirrhosis, liver cirrhosis-related complications, subjects with HBsAg seroclearance, subjects with HBV DNA <15 IU/mL, Serial changes of liver stiffness assessed by Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, PhD, Principal Investigator — Asan Medical Center
Locations (10):
- South Korea (10):
  - Kyungpook National University Hospital, Daegu
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung-Hee University Hospital, Seoul
  - Samsung Medical center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No